CLINICAL TRIAL: NCT06049472
Title: Exploring Patient Engagement Patterns and Participation Trends in Mantle Cell Lymphoma Clinical Trials
Brief Title: Patient Perspectives in Mantle Cell Lymphoma Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 70247036
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical studies with a distinct emphasis on mantle cell lymphoma play a pivotal role in evaluating the safety and effectiveness of novel treatments for this disease. These trials are instrumental in ascertaining whether new medications surpass conventional therapies, providing substantial evidence to endorse their broad utilization.

This particular study stands out as it centers on the firsthand experiences of individuals battling mantle cell lymphoma who are actively engaged in a clinical trial featuring medicinal interventions. The primary objective is to meticulously scrutinize trial completion rates and voluntary withdrawals within this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mantle cell lymphoma
* No serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Concurrent participation in another therapeutic clinical trial.
* Subject has an uncontrolled infection
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mantle cell lymphoma patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a mantle cell lymphoma clinical study | 3 months
Rate of patients who remain in a mantle cell lymphoma clinical study to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nickenig C, Dreyling M, Hoster E, Pfreundschuh M, Trumper L, Reiser M, Wandt H, Lengfelder E, Unterhalt M, Hiddemann W; German Low-Grade Lymphoma Study Group. Combined cyclophosphamide, vincristine, doxorubicin, and prednisone (CHOP) improves response rates but not survival and has lower hematologic toxicity compared with combined mitoxantrone, chlorambucil, and prednisone (MCP) in follicular and mantle cell lymphomas: results of a prospective randomized trial of the German Low-Grade Lymphoma Study Group. Cancer. 2006 Sep 1;107(5):1014-22. doi: 10.1002/cncr.22093. PMID 16878325
- [Background] Campbell J, Hurtado S, Kutz C, Soto K, Ernst D. [Cytarabine and hematopoietic cell transplantation for mantle cell lymphoma. Analysis of 20 patients]. Rev Med Chil. 2019;147(1):9-17. doi: 10.4067/S0034-98872019000100009. Spanish. PMID 30848759
- [Background] Dasappa L, Suresh Babu MC, Sirsath NT, Suresh TM, Govind Babu K, Sathyanarayna V, Lokesh KN, Lakshmaiah KC. Primary gastrointestinal mantle cell lymphoma: a retrospective study. J Gastrointest Cancer. 2014 Dec;45(4):481-6. doi: 10.1007/s12029-014-9655-2. PMID 25316096

DOCUMENTS (1):
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT06049472/ICF_000.pdf